CLINICAL TRIAL: NCT01790841
Title: Master Study of the BIOTRONIK DF4 System
Brief Title: DF4 Master Study (Safety and Efficacy Study)
Status: Completed | Type: Observational
Sponsor: Biotronik SE & Co. KG (Industry)
Responsible Party: Sponsor
Other Study IDs: 54
Record Dates: First submitted 2013-02-12; First posted 2013-02-13 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-04

CONDITIONS: Ventricular Tachycardia; Ventricular Fibrillation; Sudden Cardiac Death; Heart Failure
MeSH Terms: conditions — Tachycardia, Ventricular; Ventricular Fibrillation; Death, Sudden, Cardiac; Heart Failure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ICD system with DF4 connection: Iforia/Ilesto ICD with DF4 connection and Linox smart DF4 lead/ Protego
  Interventions: Device: Iforia/Ilesto ICD/CRT-D, Linox smart DF4 lead/ Protego
- ICD system with DF-1 connection: Ilesto/Iforia ICD with DF-1 connection
  Interventions: Device: Iforia/Ilesto ICD/CRT-D, Linox smart DF4 lead/ Protego

INTERVENTIONS:
Device: Iforia/Ilesto ICD/CRT-D, Linox smart DF4 lead/ Protego

SUMMARY:
The purpose of the study is to proof the safety and efficacy of the new ICD sytem (Iforia/Ilesto). The devices are available with DF-1 and DF4 connection. A special focus is set on the ICD system with DF4 connection.

ELIGIBILITY:
Inclusion Criteria:

* Patient has provided written informed consent.
* Patient has standard ICD/CRT-D indication.
* Patient accepts Home Monitoring concept.
* Patient is able to attend the planned hospital follow-up visits.
* Patient has legal capacity and ability to consent.

Exclusion Criteria:

* Patient has a standard contra-indication for ICD/CRT-D therapy.
* Age < 18 years
* Patient is pregnant or breastfeeding.
* Patient is expected to receive ventricular assist device or heart transplantation within the next 12 months.
* Life expectancy of less than 12 months.
* Participating in any other clinical study of an investigational cardiac drug or device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with standard ICD/CRT-D indication who are referred to the hospital.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2013-02; Primary Completion 2015-05 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Serious adverse device effect (SADE) rate related to the ICD with DF4 connection | until 3 month follow-up
SADE rate related to the Linox smart DF4 lead (ICD shock lead) | until 3 month follow-up
Shift rate of the painless shock impedance measurement | between 3 and 6 month follow-up
Pacing threshold comparison between Linox smart DF-1 and Linox smart DF4 lead | 3 month follow-up

SECONDARY OUTCOMES:
Comparison of automatic atrial pacing threshold test vs. manual measurement | 3 month follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Universitaetsmedizin Greifswald, Greifswald, Germany